CLINICAL TRIAL: NCT06777602
Title: An Open-label Phase 1 IV Study to Evaluate Metabolism, Excretion, and Mass Balance of [14C]MK-5475 in Healthy Participants
Brief Title: A Clinical Study To Understand How Radiolabeled MK-5475 Is Taken Up By The Body, Broken Down And Then Removed From The Body in Healthy Participants (MK-5475-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5475-011; MK-5475-011 (Other: MSD)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] MK-5475 (Experimental): [14C] MK-5475 is administered as single IV bolus dose of 100μg on Day 1.
  Interventions: Drug: [14C] MK-5475

INTERVENTIONS:
Drug: [14C] MK-5475 — [14C] MK-5475 is administered as a single IV bolus dose in healthy male participants on Day 1.

SUMMARY:
The goal of this study is to understand how radiolabeled MK-5475 administered intravenously (IV) is taken up by the body, broken down and then removed from the body in healthy male participants. The study also aims to understand how much of the compound is broken down and how much leaves the body unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health.
* Body mass index (BMI) >18 and ≤32 kg/m2, inclusive.

Exclusion Criteria:

* Has history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
* Has had a major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) or blood products within 4 weeks prior to the prestudy (screening).
* Has history of exposure to significant diagnostic or therapeutic radiation or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
* Has participated in more than 3 radiolabeled drug studies in the last 12 months.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult male participants
Enrollment: 8 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Amount Excreted in Urine (Aeu) | At designated time points (Up to ~ 23 days)
  Amount of [14C]MK-5475 and its metabolites excreted in urine (Aeu) derived from urine collections at each sampling interval.
Cumulative Aeu | At designated time points (Up to ~ 23 days)
  Cumulative amount of [14C] MK-5475 and its metabolites excreted in urine derived from urine collections at each sampling interval
Percentage Excreted in Urine (feu) | At designated time points (Up to ~ 23 days)
  Percentage of [14C]MK-5475 and its metabolites excreted in urine derived from urine collections at each sampling interval.
Cumulative feu | At designated time points (Up to ~ 23 days)
  Cumulative percentage of [14C]MK-5475 and its metabolites excreted in urine derived from urine collections at each sampling interval.
Amount Excreted in Feces (Aef) | At designated time points (Up to ~ 23 days)
  Amount of [14C]MK-5475 and its metabolites excreted in feces derived from feces collections at each sampling interval.
Cumulative Aef | At designated time points (Up to ~ 23 days)
  Cumulative amount of [14C]MK-5475 and its metabolites excreted in feces derived from feces collections at each sampling interval.
Cumulative Fef | At designated time points (Up to ~ 23 days)
  Cumulative percentage of [14C]MK-5475 and its metabolites excreted in feces derived from feces collections at each sampling interval.
AUC0-t | At designated time points (Up to ~ 23 days)
  Area under concentration time curve (AUC) from time zero to the last quantifiable concentration derived from the whole blood and plasma concentration-time profiles following IV administration of [14C]MK-5475.
AUC0-infinity | At designated time points (Up to ~ 23 days)
  AUC from time zero extrapolated to infinity derived from the whole blood and plasma concentration-time profiles following IV administration of [14C]MK-5475.
Maximum Plasma Concentration (Cmax) | At designated time points (Up to ~ 23 days)
  Cmax is the measure of the maximum amount of [14C]MK-5475 in the plasma after the dose is given.
Half-life t1/2 | At designated time points (Up to ~ 23 days)
  T1/2 is the time required for [14C]MK-5475 concentration in the plasma to decrease by 50%.
Time to Maximum Plasma Concentration (Tmax), | At designated time points (Up to ~ 23 days)
  Tmax is a measure of the time to reach the maximum concentration in the plasma after the [14C]MK-5475 dose.
Apparent Total Clearance (CL; MK-5475 only) | At designated time points (Up to ~ 23 days)
  CL is defined as apparent total clearance of [14C]MK-5475 from plasma after IV administration
Apparent Volume of Distribution (Vz; MK-5475 only) | At designated time points (Up to ~ 23 days)
  Vz is defined as apparent volume of distribution of [14C]MK-5475 during terminal phase after IV administration.
AUC0-infinity Plasma [14C]MK-5475/Total Radioactivity Ratio | At designated time points (Up to ~ 23 days)
  AUC time zero to infinity (0-∞) of [14C]MK-5475 in plasma/AUC0-∞ of total radioactivity in plasma.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to ~ 30 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to ~ 30 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Labcorp Clinical Research Unit Inc. (Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Menzel K, Liang Y, Chen B, Li D, Cislak D, Bajwa EK. An Intravenous Study with the Radiolabeled sGC Stimulator Frespaciguat to Assess PK, Metabolism, and Mass Balance. J Clin Pharmacol. 2025 Nov;65(11):1561-1567. doi: 10.1002/jcph.70066. Epub 2025 Jun 19. PMID 40534306
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com